CLINICAL TRIAL: NCT02973256
Title: Postoperative Oncological Care for Patients With Meningioma With Malignant Components
Brief Title: Oncological Care for Patients With Meningioma
Acronym: ATYPICMENING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: UF9759
Record Dates: First submitted 2016-10-17; First posted 2016-11-25 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Atypical Meningioma; Clear-cell Meningioma; Chordoid Meningioma; Anaplastic Meningioma; Rhabdoid Meningioma; Papillary Meningioma
Keywords: Meningioma grade II; Meningioma grade III
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Meningiomas with malignant components include grade II meningiomas (GIIM, the most common ones) and grade III meningiomas (GIIIM). They represent 5-35% of all meningiomas. Histological diagnosis of GIIM criteria were changed in 2007 and might be viewed by some as being quite subjective. "Standards of care" and consensus do not exist for GIIM, particularly in regards to performing, or not, radiotherapy after surgery. One other limitation in the literature is lack of data on health-related quality of life (HRQoL). Clinical trials for GIIM are very difficult to conduct. No results have been made available. Here, we propose to study clinical, pathological, radiological and therapeutic factors of an exhaustive population of GIIM and GIIIM patients, at national level. The main objective (for GIIM) is to assess the impact of postoperative radiotherapy, or the absence of postoperative radiotherapy, on overall survival and on quality of life

DETAILED DESCRIPTION:
Meningiomas with malignant components include grade II meningiomas (GIIM, the most common ones) and grade III meningiomas (GIIIM). They represent 5-35% of all meningiomas. Histological diagnosis of GIIM criteria were changed in 2007 and might be viewed by some as being quite subjective. "Standards of care" and consensus do not exist for GIIM, particularly in regards to performing, or not, radiotherapy after surgery. One other limitation in the literature is lack of data on health-related quality of life (HRQoL). Clinical trials for GIIM are very difficult to conduct. No results have been made available.

Main objective: to assess the impact of postoperative radiotherapy after GIIM surgery on overall survival (OS) in a population-setting study.

Secondary objectives (for GIIM and GIIIM):

* Evaluate the recurrence/progression free survival (PFS), volumetric velocity of the tumor growth (VVTG) after surgery and other treatment.
* Evaluate long term HRQoL.
* Evaluate the relevance and impact of histopathological review in a population setting.
* Looking for prognostic (clinical, radiological and biological) factors.
* Proposing therapeutic decision trees in general or for certain categories of patients.
* Identifying relevant cases to conduct further studies to identify new therapeutic targets.
* Perspectives for the TUCERA network to help design specific prospective projects.
* Looking for disparities in care management, survival and HRQoL in the various regions of France.

Design of the study: nationwide population-based study analysis and patterns of care/quality of care study, for all cases of incident GIIM and GIIIM operated in Metropolitan France during the 2007-2010 period.

The methodology used is based on a multidisciplinary national network already established by the French Brain Tumor DataBase (FBTDB), with the active participation of societies involved in the French neuro-oncology and the "Inter Groupe Coopérateur en Neuro-Oncologie", labeled by the French National Cancer Institute.

The FBTDB has already identified all incident cases of GIIM (n=1046) and GIIIM (n=158) operated in Metropolitan France from 2007 to 2010.

The study proposed is a retrospective study based on the medical charts of all these patients.

Furthermore, for all surviving patients not lost to follow-up, the follow-up consultations will include a prospective HRQoL evaluation (cutoff date: 2019/11/30).

It will be conducted a systematic pathological review (with eventually additional biological work-up), and a study of prognostic factors (clinical, radiological, biological), treatments administered, OS, PFS.

Primary endpoint: OS. The statistical analysis (to answer to the main question) will concern all GIIM only.

Hypothesis:

Experimental group: Group of GIIM with postoperative radiotherapy (n=314). Control group: Group of GIIM with postoperative follow-up only (n=732). With a bilateral type I error of 5% (two-sided) and a statistical power of 80% we will be able to demonstrate that postoperative radiotherapy will be associated with a Hazard ratio (mortality risk) of 0.80.

Secondary endpoints (for GIIM and GIIIM):

* PFS, VVTG after surgery and other treatment.
* HRQoL will be assessed using EORTC QLQ-C30, BN20 questionnaires, Europol EQ5D, and with a questionnaire on professional and social activities (HRQoL will be assessed for all patients alive, every six months, since inclusion, for an 18-month period).
* Mapping between HRQoL questionnaires.
* Concordance/discordance analysis between the initial histological diagnosis and the diagnosis of the pathological review.
* Conduct an inventory of cryopreserved material available for translational research.

It is expected to:

* Define subgroups of patients, according to prognostic factors, which would benefit from postoperative radiotherapy in GIIM.
* Define subgroups of patients, according to their prognostic factors, which would benefit from not having postoperative radiotherapy in GIIM.
* Propose personalized therapeutic attitudes according to prognostic factors (clinical, radiological, and biological) in general, but also for specific categories of patients such as elderly subjects.
* Define subgroups of GIIM and GIIIM that will justify conducting trials in the framework of the TUCERA network.
* Evaluate in population settings, the relevance and impact of a systematic histopathological review.
* Develop HRQoL evaluation in population settings.
* Acquire better knowledge of prognostic factors (clinical, radiological and biological) for GIIM and GIIIM, their natural history, and maybe help determine elements able to differentiate GIIM that will progress to GIIIM, from those that will remain GIIM.
* Build a clinical-biological database to identify and/or develop new therapeutic targets in GIIM and GIIIM.
* Evaluate potential disparities in terms of survival and HRQoL in the different French regions, and if some disparities are found, look for eventual causes.

ELIGIBILITY:
Inclusion Criteria :Patient with a GIIM incident (atypical, chordidic and clear cell meningiomas) and GIIIM (anaplastic, papillary and rhabdoid meningiomas) operated in metropolitan France during the period 2007-2010

Exclusion Criteria :

* Patient with GIM
* Non-operated meningioma patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a histological diagnosis of GIIM and GIIIM in metropolitan France
Sampling Method: Non-Probability Sample
Enrollment: 1204 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 10 years, since diagnosis
  Description: Assessing the impact of postoperative radiotherapy after surgery on overall survival (OS) in population-based study of GIIM patients. Overall survival, the primary endpoint of this study, is defined as the time from surgery (histological diagnosis) to the time of death from any cause. Alive Patients at the time of the final analysis or who became lost to follow-up will be censored at their last date of giving news

SECONDARY OUTCOMES:
the tumor growth | up to 10 years, since diagnosis
  The tumor growth after surgery and other treatment (based on successive MRIs) will be determined by the volumetric velocity of the tumor growth (mm3/year)
Progression/Recurrence Free Survival, will be measured by month | up to 10 years, since diagnosis

OTHER OUTCOMES:
Evaluation of the quality of life | baseline, 6 months, 12 months 18 months
  Change from baseline in patients with a I and II grade glioma, defined by quality-of-life parameters Health related Quality of Life will be assessed using EORTC QlQ C30 and BN 20 questionnaires, Europol EQ5D, and a specific questionnaire on professional and social activities.
  -EORTC QLQ-C30: Score at baseline, The change in the EORTC QLQ-C30 score from baseline to endpoint
  -EORTC QLQ-BN20: Score at baseline, The change in the EORTC QLQ-C30 score from baseline to endpoint
  * Europol EQ5D Score at baseline, The change in the EORTC QLQ-C30 score from baseline to endpoint
  * Specific questionnaire on professional and social activities:
  Score at baseline, The change in the Specific questionnaire on professional and social activities score from baseline to endpoint
diagnosis of the central pathological review. | 1 day
  Concordance/discordance analysis between the initial histological diagnosis and the diagnosis of the central pathological review.

CONTACTS AND LOCATIONS:
Overall Officials: LUC BAUCHET, MD, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided